CLINICAL TRIAL: NCT06794567
Title: Improving Diagnosis for Genetic Kidney Disease Through Early Genomic Assessment
Brief Title: Genomic First Testing in Chronic Kidney Disease
Status: Not yet recruiting | Type: Observational
Sponsor: Dervla Connaughton (Other)
Collaborators: London Health Sciences Centre (Other); London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor-Investigator, Dervla Connaughton, Principal Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Organization: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Other Study IDs: Genomic First Testing in CKD
Record Dates: First submitted 2025-01-08; First posted 2025-01-27 (Actual); Last update posted 2025-01-27 (Actual); Status verified 2025-01

CONDITIONS: Chronic Kidney Disease(CKD); Genetic Kidney Disease
Keywords: Chronic Kidney Disease; Genetic Testing; Genome wide sequencing
MeSH Terms: conditions — Renal Insufficiency, Chronic | interventions — Genetic Testing

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — DNA extracted from blood and saliva samples.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- < 1 year since diagnosis of kidney disease
  Interventions: Diagnostic Test: Genetic Testing
- > 1 year since diagnosis of kidney disease
  Interventions: Diagnostic Test: Genetic Testing

INTERVENTIONS:
Diagnostic Test: Genetic Testing — Early access to genetic testing.

SUMMARY:
This multi-center study examines the role of genetic testing in patients with chronic kidney disease (CKD) who are identified as being at risk for genetic kidney disease, based on Ontario Health's Provincial Genetic Program (OH-PGP) guidelines. Participants will be assigned to either genome-wide sequencing or standard genetic testing, depending on when they were initially diagnosed with kidney disease.

To evaluate the impact of genetic testing, patients and caregivers will complete quality-of-life questionnaires before and after testing. Participants may also choose to take part in a one-on-one interview at the end of the study to provide additional insights. They will have the option to link their data to the Institute for Clinical Evaluative Sciences (ICES), allowing researchers to explore health outcomes such as the costs of genetic testing and healthcare resource use.

Family members of participants will be invited to provide DNA samples to help identify genetic changes in the affected individual. Referring physicians will complete a survey to assess the clinical value of genetic testing for each patient they refer. We will perform an economic analysis comparing the genome wide sequencing to the standard genetic testing group.

The study's findings will offer important guidance on how genetic testing influences patient care, clinical outcomes, and the timing of genomic assessments in managing CKD.

DETAILED DESCRIPTION:
This multi-center study examines the role of genetic testing in patients with chronic kidney disease (CKD) who are identified as being at risk for genetic kidney disease, based on Ontario Health's Provincial Genetic Program (OH-PGP) guidelines. Participants will be assigned to either genome-wide sequencing or standard genetic testing, depending on when they were initially diagnosed with kidney disease.

To evaluate the impact of genetic testing, patients and caregivers will complete quality-of-life questionnaires before and after testing. Participants may also choose to take part in a one-on-one interview at the end of the study to provide additional insights. They will have the option to link their data to the Institute for Clinical Evaluative Sciences (ICES), allowing researchers to explore health outcomes such as the costs of genetic testing and healthcare resource use.

Family members of participants will be invited to provide DNA samples to help identify genetic changes in the affected individual. Referring physicians will complete a survey to assess the clinical value of genetic testing for each patient they refer. We will perform an economic analysis comparing the genome wide sequencing to the standard genetic testing group.

The study's findings will offer important guidance on how genetic testing influences patient care, clinical outcomes, and the timing of genomic assessments in managing CKD.

ELIGIBILITY:
Patients:

Inclusion Criteria:

1. A diagnosis of CKD warranting a referral to a nephrologist for further assessment AND
2. Screen positive for potential genetic kidney disease using the Ontario Health Provincial Genetics Program Eligibility Criteria for genetic assessment in CKD AND
3. Index participant or substitute decision maker (SDM) can provide informed consent to participate.

Exclusion Criteria:

1. Participant or SDM is unable to provide consent, for any reason, to be an unsuitable candidate for the study.
2. Fail screening as set out by the Provincial Genetics Program Eligibility Criteria for genetic assessment in CKD.

Family Members:

Inclusion Criteria:

1. Family/caregiver or SDM can provide informed consent to participate AND
2. Related patient participant must be enrolled in the study.

Exclusion Criteria:

1. Family/caregiver or SDM is unable to provide consent, for any reason, to be an unsuitable candidate for the study.
2. Related patient participant is not enrolled in the study.

Healthcare Provider:

Inclusion Criteria 1. Provided a referral for at least one study participant.

Exclusion Criteria:

1. Is not a referring healthcare provider.

Qualitative Sub-Study:

Inclusion Criteria:

1. Patient participant who is enrolled in the main study.
2. 18 years or older.
3. The guardian for a minor

Exclusion Criteria:

1. <18 years of age unless the guardian can conduct the interview
2. Patient participant who is not enrolled in the main study.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients, Family Members, Healthcare providers
Sampling Method: Non-Probability Sample
Enrollment: 2400 (Estimated)
Dates: Start 2025-03-01 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic yield and time to diagnosis | Study duration
  Our primary outcome is to address the need for high diagnostic yields and short times to diagnosis for chronic kidney disease as highlighted by our patient partner board by comparing a genome-wide sequencing approach to the standard genetic testing in patients at risk of genetic kidney disease

CONTACTS AND LOCATIONS:
Locations (1):
- London Health Sciences Centre, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No